CLINICAL TRIAL: NCT00594737
Title: An Open Label Pilot Study of the Effects of Memantine Administration on FDG-PET in Frontotemporal Dementia
Brief Title: Open Label Pilot Study of the Effects of Memantine on FDG-PET in Frontotemporal Dementia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tiffany Chow, MD (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor-Investigator, Tiffany Chow, MD, Senior Scientist, Assoc. Prof. University of Toronto, Rotman Research Institute at Baycrest
Organization: Rotman Research Institute at Baycrest (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Baycrest.Ebixa.FTD-001; Lundbeck 11627A
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-06

CONDITIONS: Frontotemporal Dementia
Keywords: PET; frontotemporal dementia; memantine; Pick's disease
MeSH Terms: conditions — Frontotemporal Dementia; Pick Disease of the Brain | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: memantine hydrochloride — memantine hydrochloride oral tablets, 10mg po bid
  Other Names: Ebixa; Namenda

SUMMARY:
Memantine has been approved for use in Alzheimer's disease. Its mechanism of action raises questions of whether it can also be effective for non-Alzheimer's dementias such as frontotemporal dementia (FTD), which currently has no disease-modifying treatment.

This is an open-label study to probe the effects of memantine in 15 outpatients diagnosed with FTD, as shown objectively by comparing PET scans performed before and after use of the medication. The specific type of PET scan, FDG-PET, allows the investigators to gauge the effects of memantine on cortical activity levels. The investigators hypothesize that subjects on memantine will show normalization of cortical metabolic activity.

ELIGIBILITY:
Inclusion Criteria:

* Must meet criteria for frontotemporal lobar degeneration (FTD) by Neary et al. criteria. 28 Subjects may have either the behavioural or the aphasic variant of FTD.
* Able to undergo psychometric testing.
* Must have reliable informant with daily contact with patient
* May be taking concurrent psychotropic medications, but must be on stable dosing regimen for 3 months prior to trial enrollment
* On the basis of a physical examination, medical history (including psychiatric and neurological), and results of blood chemistry carried out at screening visit, the patient in the investigator's opinion is considered healthy.
* Signed Informed Consent must be obtained from the patient or legally responsible representative and the informant prior to initiating any study specific procedures.

Exclusion Criteria:

* Complaint of recurrent or persistent dizziness or constipation
* Abnormal chemistry panel particular with respect to ruling out renal insufficiency or failure. We will exclude those patients with creatinine clearance (CLcr) < 50ml/min, per the Sakana equations for men and women.
* Angina, myocardial infarction, severe hypertension, severe cardiac arrhythmia, unstable diabetes mellitus, or new abnormalities on EKG within the past year.
* Any current malignancy, or any clinically significant hematological, endocrine, renal, hepatic, gastrointestinal or non-dementia neurological disease. If the condition has been stable for at least the past year and is judged by the investigators not to interfere with the patient's participation in the study, the patient may be included. Basal cell carcinoma is an exception.
* Non-English speaking, as cognitive tests will be in English.
* Evidence of other neurological or psychiatric disorders which preclude diagnosis of FTD (including, but not limited to, stroke, Parkinson's disease, any psychotic disorder, severe bipolar or unipolar depression) within the past year
* Current or prior history of uncontrolled seizure disorder, due to seizures reported as adverse events with memantine.
* Patients with suspected alcohol or substance abuse within last 1 year. If past history of abuse or dependence must have been abstinent for 1 year with continuing progression of dementia despite abstinence.
* Patients with active delusions or hallucinations at the time of screening.
* Female patients who are not at least two years post-menopausal or surgically sterile. Pre-menopausal women will be excluded; because almost all women are post-menopausal at the age of onset of FTD, we do not anticipate having to exclude more than one potential subject on the basis of this one exclusion criterion.
* Use of investigational drugs or participation in another investigational drug study within 3 months of screening.
* Patients who have previously been treated with memantine or have participated in an investigational study with memantine.
* Patients with history of severe drug allergy or hypersensitivity or known hypersensitivity to amantadine or memantine.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Metabolic activity in frontal and temporal lobes. | 6 months

SECONDARY OUTCOMES:
Behavioural inventories, UPDRS Motor scale. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany W Chow, MD, Principal Investigator — Rotman Research Institute at Baycrest, University of Toronto
Locations (1):
- Baycrest, Toronto, Ontario, Canada

REFERENCES:
- [Background] Swanberg MM. Memantine for behavioral disturbances in frontotemporal dementia: a case series. Alzheimer Dis Assoc Disord. 2007 Apr-Jun;21(2):164-6. doi: 10.1097/WAD.0b013e318047df5d. PMID 17545743
- [Result] Chow TW, Binns MA, Freedman M, Pollock BG, Verhoeff NPG, Graff-Guerrero A. Pre- and post-memantine FDG-PET imaging in frontotemporal dementia. Am J Geriatr Psychiatry 2009;17(3 Supp 1): A73.
- [Result] Chow TW, Graff-Guerrero A, Verhoeff NP, Binns MA, Tang-Wai DF, Freedman M, Masellis M, Black SE, Wilson AA, Houle S, Pollock BG. Open-label study of the short-term effects of memantine on FDG-PET in frontotemporal dementia. Neuropsychiatr Dis Treat. 2011;7:415-24. doi: 10.2147/NDT.S22635. Epub 2011 Jul 13. PMID 21792308
- [Result] Chow TW, Fam D, Graff-Guerrero A, Verhoeff NP, Tang-Wai DF, Masellis M, Black SE, Wilson AA, Houle S, Pollock BG. Fluorodeoxyglucose positron emission tomography in semantic dementia after 6 months of memantine: an open-label pilot study. Int J Geriatr Psychiatry. 2013 Mar;28(3):319-25. doi: 10.1002/gps.3832. Epub 2012 Jun 4. PMID 22674572
- See also: PET Imaging Centre website — http://www.camhpet.ca/
- See also: Association for Frontotemporal Dementias — http://www.theaftd.org